CLINICAL TRIAL: NCT07339436
Title: Effect of Lower Body Plyometric Training on Neuromuscular Adaptations, Hormonal Factors, Functional Performance, and Upper Body Muscle Thickness in Basketball Players
Brief Title: Lower Body Plyometric Training Effects on Upper Body in Basketball Players
Acronym: LBPT-VST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birjand University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohsen mohammadnia ahmadi, Assistant Professor, Department of Sport Sciences, Faculty of Sport Sciences, University of Birjand, Birjand University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Birjand-Plyometric-1403; IR.BIRJAND.REC.1403.016 (Other: Research Ethics Committees of University of Birjand)
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Basketball Performance
Keywords: plyometric training; neuromuscular adaptation; hormonal factors; cross-education
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined Lower-Upper Body Plyometric Training (LUBPT) - n=17 (Experimental): Combined Lower-Upper Body Plyometric Training (LUBPT) group received an 8-week plyometric program targeting both lower and upper body, 3 sessions per week (total 24 sessions). Lower body exercises included hurdle jumps (40-60 cm height) and depth jumps (from 40 cm box). Upper body exercises consisted of dynamic push-ups. Progression: Weeks 1-2 (sessions 1-6): 2 sets of 8 reps per exercise; Weeks 3-4 (sessions 7-12): 3 sets of 10 reps; Weeks 5-6 (sessions 13-18): 3 sets of 12 reps; Weeks 7-8 (sessions 19-24): 4 sets of 15 reps. Rest intervals: 60-90 seconds between sets, 3 minutes between exercises. Training was performed in addition to regular basketball practice. Pre- and post-tests assessed neuromuscular adaptations (EMG: pectoralis major, rectus abdominis, triceps brachii), hormonal factors (growth hormone, testosterone), muscle thickness (biceps brachii, pectoralis major via ultrasound elastography), and functional performance (overhead medicine ball throw, Sargent jump height/pow
  Interventions: Behavioral: Plyometric Training
- Upper Body Plyometric Training (UBPT, n=18) (Experimental): Upper Body Plyometric Training (UBPT) group received an 8-week plyometric program targeting only upper body, 3 sessions per week (total 24 sessions). Primary exercise: dynamic push-ups. Progression: Weeks 1-2 (sessions 1-6): 2 sets of 8 reps; Weeks 3-4 (sessions 7-12): 3 sets of 10 reps; Weeks 5-6 (sessions 13-18): 3 sets of 12 reps; Weeks 7-8 (sessions 19-24): 4 sets of 15 reps. Rest intervals: 60-90 seconds between sets. Lower body training was not included; participants continued regular basketball practice. Assessments pre- and post-intervention: serum growth hormone and testosterone levels; muscle thickness of biceps brachii and pectoralis major (ultrasound elastography); EMG activity (RMS) of anterior brachii, pectoralis major, quadriceps femoris, rectus abdominis, triceps brachii; functional tests including overhead medicine ball throw distance, Sargent jump (height and power), and standing long jump.
  Interventions: Behavioral: Plyometric Training
- Control (CON, n=15) (No Intervention): Control (CON) group did not receive any plyometric training intervention. Participants continued their regular basketball training routine (technical/tactical drills, scrimmages) for 8 weeks, 3-5 sessions per week, without additional structured plyometric exercises for lower or upper body. No changes to standard practice schedule. This group served as the non-intervention comparator to assess the specific effects of plyometric training. Pre- and post-assessments (48-72 hours before start and after week 8) included: hormonal measurements (serum growth hormone and testosterone via ELISA); muscle thickness (right/left biceps brachii and pectoralis major using ultrasound elastography); neuromuscular electrical activity (surface EMG RMS during standardized tasks for anterior brachii, pectoralis major, quadriceps femoris, rectus abdominis, triceps brachii); physical performance tests (overhead medicine ball throw distance in meters, Sargent vertical jump height and power in kg m/s, standing

INTERVENTIONS:
Behavioral: Plyometric Training — 8-week plyometric training program, 3 sessions per week. Lower body exercises: hurdle jumps (40-60 cm) and depth jumps (from 40 cm box). Upper body exercises: dynamic push-ups. Progression: increasing sets (2-4) and repetitions (8-15) over 8 weeks. Rest: 60-90 seconds between sets, 3 minutes between exercises. Administered in addition to regular basketball training.
  Arms: Combined Lower-Upper Body Plyometric Training (LUBPT) - n=17; Upper Body Plyometric Training (UBPT, n=18)

SUMMARY:
The present study investigates effect of lower body plyometric training on upper body performance, muscle size, hormonal factors, and neuromuscular activity in male basketball players, with a focus on vertical strength transfer (VST). In this semi-experimental study, 50 male basketball players (aged 16-18 years, with at least 2 years of experience) were randomly divided into three groups: combined lower-upper body plyometric training (LUBPT), upper body training (UBPT), and control (CON). The 8-week training program, 3 sessions per week, included hurdle jumps, depth jumps, and dynamic push-ups. Assessments included serum levels of growth hormone and testosterone, muscle thickness (elastography), muscle electrical activity (EMG), and sports performance (overhead medicine ball throw, Sargent jump, long jump) in pre- and post-tests.

DETAILED DESCRIPTION:
This semi-experimental study was conducted to investigate the effects of an 8-week lower body plyometric training program on neuromuscular adaptations, hormonal factors, functional performance, and upper body muscle thickness in male basketball players, with a focus on vertical strength transfer (VST).

Fifty male basketball players aged 16-18 years with at least 2 years of competitive experience were recruited and randomly allocated into three groups: Combined Lower-Upper Body Plyometric Training (LUBPT, n=17), Upper Body Plyometric Training only (UBPT, n=18), and Control (CON, n=15). The control group continued regular basketball training without additional plyometric exercises.

The intervention lasted 8 weeks with 3 sessions per week. The plyometric program consisted of lower body exercises (hurdle jumps at 40-60 cm height and depth jumps from a 40 cm box) and upper body exercises (dynamic push-ups). Training volume and intensity progressed gradually over the 8 weeks (sessions 1-8: 2-3 sets of 8-10 repetitions; sessions 9-16: 3-4 sets of 10-12 repetitions; sessions 17-24: 4 sets of 12-15 repetitions), with 60-90 seconds rest between sets and 3 minutes between exercises.

Pre- and post-intervention assessments included:

* Serum levels of growth hormone and testosterone (blood samples taken in fasting state).
* Upper body muscle thickness (biceps brachii and pectoralis major) measured using ultrasound elastography.
* Neuromuscular activity (root mean square, RMS) of anterior brachii, pectoralis major, quadriceps femoris, rectus abdominis, and triceps brachii muscles using surface electromyography (EMG) during standardized movements.
* Functional performance tests: overhead medicine ball throw, Sargent vertical jump (height and power), and standing long jump.

All measurements were performed 48-72 hours before the start of training and 48-72 hours after the final training session. Statistical analysis was conducted using ANOVA with significance set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Male basketball players with at least 2 years experience

Exclusion Criteria:

* injury

Ages: 16 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — male basketball players
Enrollment: 50 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Overhead medicine ball throw | Baseline and after 8 weeks
  Participants stood with feet shoulder-width apart, holding a 2 kg medicine ball at the abdomen with both hands, then brought the ball behind the head with slight knee bend, and performed an explosive and strong throw forward with full force. The distance was measured with a tape measure and considered as overhead medicine ball throw performance [22]. In the above test, electrical activity of pectoralis major, rectus abdominis, quadriceps femoris, Anterior Brachii, and triceps brachii muscles was recorded.
Overhead medicine ball throw | pre and post intervention
  Participants stood with feet shoulder-width apart, holding a 2 kg medicine ball at the abdomen with both hands, then brought the ball behind the head with slight knee bend, and performed an explosive and strong throw forward with full force. The distance was measured with a tape measure and considered as overhead medicine ball throw performance [22]. In the above test, electrical activity of pectoralis major, rectus abdominis, quadriceps femoris, Anterior Brachii, and triceps brachii muscles was recorded.

SECONDARY OUTCOMES:
Growth hormone | Baseline and after 8 weeks
  For blood sampling, participants were asked to avoid sports activity for at least 48 hours before the test and attend the laboratory between 8-9 AM after 12 hours of fasting. Blood was drawn in a sitting position from the antecubital vein of volunteers in 6 ml amounts by a laboratory expert and collected in test tubes. Then, it was centrifuged for 10 minutes at 5000 rpm, and the separated serum was transferred to microtubes and stored in a -20°C freezer for analysis. Post-test blood sampling was the same as pre-test and 48 hours after the last training session. The highly accurate electrochemiluminescence (ECLIA) method and Siemens IMMULITE 2000 XPi Immunoassay System device with Siemens-specific kits with 0.0001 mIU/L accuracy were used to examine changes in growth hormone and testosterone levels of participants

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sport Sciences, University of Birjand, Birjand, South Khorasan Province, Iran

IPD SHARING:
Plan to Share IPD: No